CLINICAL TRIAL: NCT03857113
Title: 99mTechnetium Based PSMA-Radioguided Assisted Surgery for Prostate Cancer (TRACE) Feasibility Study
Brief Title: Technetium Based Radioguided Surgery for Prostate Cancer (TRACE) Study
Acronym: TRACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: M19TRA
Record Dates: First submitted 2018-11-19; First posted 2019-02-27 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PSMA-radioguided surgery: Tc-99m-PSMA combined with a gamma probe, guidance of the surgical resection of recurrent PC lymph node metastases
  Interventions: Procedure: PSMA-radioguided surgery

INTERVENTIONS:
Procedure: PSMA-radioguided surgery — PSMA-radioguided surgery

SUMMARY:
PSMA-radioguided surgery

DETAILED DESCRIPTION:
Given the difficulty visualizing lymph node involvement with pre-operative imaging alone, and the potential to miss metastatic nodal involvement on template PLND, radioguided surgery has been proposed as a technique to improve intra-operative detection and clearance. 99mTechnetium (99mTc) is a frequently used radioisotope in nuclear medicine, with favourable radiation properties and commercial availability[11]. It has a 6-hour half-life, and is suited to allow target tissue accumulation, while minimizing patients and investigator radiation exposure. Novel molecule-targeted radiopharmaceuticals using 99mTC and other radioisotopes in the setting of PC have increasing potential for diagnostic imaging, monitoring of therapeutic interventions and directed surgery[11, 12]. In relation to radioguided surgery, 99mTC -based PSMA-radioguided surgery (99mTc-PSMA-RGS) was deployed in a feasibility study. Using a specifically designed 99mTc based tracer, 99mTc-mas3-y-nal-k(Sub-KuE), or in short Tc-99m-PSMA I&S, combined with a gamma probe, guidance of the surgical resection of recurrent PC lymph node metastases was undertaken in 132 patients, yielding a sensitivity of 84% and specificity of 100% and detecting metastases as small as 3mm[15, 16]. This raises the question as to whether a combination of PSMA PET/CT imaging and PSMA-radioguided surgery may increase the cure rate in patients undergoing operative management of PC, by increasing detection sensitivity and specificity of nodal metastases.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged ≥ 18 years.
* Hormone-sensitive recurrent prostate cancer after radical prostatectomy
* <3 soft tissue lesions (lymph node; connective tissue) within the pelvis or retroperitoneum with sufficient PSMA expression (≥3 times regional vascular activity level) as determined by PSMA-based PET
* PSA-value <4ng/mL
* Had a PSMA PET/CT within 60 days before surgery
* Suitable for salvage lymph node dissection, as per institutional guidelines.
* WHO performance status 0,1, or 2.
* Written informed consent.

Exclusion Criteria:

* Suspicion of local recurrent prostate cancer within the prostatic fossa not treatable by surgery
* Nonregional lymphadenopathy (cM1a) or distant metastases (cM1b/c) as assessed by preoperative PSMA PET/CT.
* Ongoing androgen deprivation therapy (ADT) or within 6 months prior to surgery.
* Severe claustrophobia interfering with PET/CT or SPECT/CT scanning.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — men with prostate cancer
Study Population: men with hormone-sensitive recurent prostate cancer
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
sensibility of 99mTc-PSMA Radioguided surgery in lymph node dissection | through study completion, an average of two days
  sensibility of 99mTc-PSMA-I&S by calculating the percentage of PSMA avid lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Pim van Leeuwen, MD, PHD, Principal Investigator — NKI-AvL
Locations (1):
- AVL, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No